CLINICAL TRIAL: NCT05195437
Title: Evolution of the Quality of Life of Short Stature Children Treated With Growth Hormone : Evaluation at Adult Size
Brief Title: Evolution of the Quality of Life of Short Statured Children Treated With Growth Hormone : Evaluation at Adult Size
Acronym: HF QoL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211523; 2024-A01272-45 (Other: IDRCB number)
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Growth Hormone Treatment
Keywords: Growth hormone treatment; Quality of Life of Short Stature Youth (QoLiSSY) questionnaire; Pediatric Quality of Life Inventory (PedsQL) 4.0; Quality of life improvement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Growth hormone treatment: Adolescents and young adults followed or having been followed by the endocrinology, gynecology and pediatric diabetology department of the Necker Enfants Malades hospital, who reached their final height and who have been treated with growth hormone due to short stature.
  Interventions: Other: QoLiSSY and PedsQL 4.0 questionnaires

INTERVENTIONS:
Other: QoLiSSY and PedsQL 4.0 questionnaires — Patients have been reaching adult size complete the two questionnaires of the study :
  Quality of Life of Short Stature Youth questionnaire (QoLiSSY), assessing health-related quality of life in short stature youth.
  Pediatric Quality of Life Inventory (PedsQL) 4.0 : general health-related quality of life.
  The patients have previously completed the PedsQL 4.0 and QoLiSSY questionnaires when starting their growth hormone therapy and after one year of growth hormone therapy.

SUMMARY:
Short stature can lead to emotional and social stress in children and adolescents, as well as their parents. Children and their parents want to be able to identify the cause of stunted growth and address it with treatment. Mitigating the impact of short stature on quality of life is one of the main goals of treatment. The quality of life in children can be measured using adapted self-questionnaires.

The investigative team published in 2019 the results of a preliminary study which shows that after one year of treatment with growth hormone, the quality of life improves in children, in particular on the scales emotional and social. These evaluations were carried out in particular thanks to the general questionnaire of quality of life: Pediatric Quality of Life Inventory (PedsQL) 4.0, but also via a specific questionnaire of the size: Quality of Life of Short Stature Youth questionnaire (QoLiSSY).

50 of the 74 patients who participated in this study have now reached their final height. The objective of the present study is to reassess this cohort using the QoLiSSY and PedsQL 4.0 questionnaires. The patient will be his own witness.

DETAILED DESCRIPTION:
Short stature can lead to emotional and social stress in children and adolescents, as well as their parents. Children and their parents want to be able to identify the cause of stunted growth and address it with treatment. Mitigating the impact of short stature on quality of life is one of the main goals of treatment. The quality of life in children can be measured using adapted self-questionnaires.

The investigative team published in 2019 the results of a preliminary study which shows that after one year of treatment with growth hormone, the quality of life improves in children, in particular on the scales emotional and social. These evaluations were carried out in particular thanks to the general questionnaire of quality of life: Pediatric Quality of Life Inventory (PedsQL) 4.0, but also via a specific questionnaire of the size: Quality of Life of Short Stature Youth questionnaire (QoLiSSY).

50 of the 74 patients who participated in this study have now reached their final height. The objective of the present study is to reassess this cohort using the QoLiSSY and PedsQL 4.0 questionnaires. The patient will be his own witness.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults followed or having been followed by the endocrinology, gynecology and pediatric diabetology department of the Necker Enfants Malades hospital and treated with growth hormone because of their short stature.
* Patient who participated in the initial study.
* Patient having reached the final height during the last consultation (growth rate less than 1 cm / year and / or bone age ≥ 15 years for girls, ≥ 17 years for boys).
* Holders of parental authority, minor patients and adult patients informed and not opposed to their participation in the study.

Exclusion Criteria:

- Refusal to participate in the study.

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and young adults followed or having been followed by the endocrinology, gynecology and pediatric diabetology department of the Necker Enfants Malades hospital, who reached their final height, who have been treated with growth hormone due to short stature and who had participed in the initial study : PedsQL 4.0 and QoLiSSY questionnaires completed at starting growth hormone therapy and after one year of growth hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Evolution of the quality of life | Day 0
  Evolution of the quality of life in short patients who have been treated with growth hormone. Comparison of the scores of the initial Quality of Life in Short Stature Youth (QoLiSSY) questionnaire (start of growth hormone treatment) compared to the scores obtained when the patients reached their final height. QoLISSY questionnaires include two different forms: parent questionnaire (children aged 4 to 18 years of age) and child questionnaire (only for children ≥8 years of age). Both questionnaires have 50 items that cover three core domains (physical, emotional, and social), and additional complementary domains. The parent questionnaire includes two additional scales (16 items) assessing parental stress and anxiety. Scores are converted in SD scores and compared to age- and gender-specific data from a reference population of children and adolescents with short stature. A total score is computed as the mean score on the three core scales.

SECONDARY OUTCOMES:
Adult-size quality of life | Day 0
  Change in scores for the two questionnaires QoLISSY and Pediatric Quality of Life Inventory (PedsQL) 4.0 at adult size.
  Children younger than 8 years of age completed the questionnaire PedsQL 4.0 with their parents. The PedsQL has 23 items that investigate physical, emotional, and social QoL, as well as school functioning. This tool has been validated in the 2- to 18-year age range. The parents complete the questionnaire if the child is younger than 5 years. After that age, the child completes the age-appropriate version of the questionnaire (5-7, 8-12, or 13-18 years). The score is expressed as a percentage, with scores from 0 to 100%, 100% being the best score. Questionnaire subscales are considered evaluable if answers are provided for at least 80% of the items. High results being associated with a better quality of life related to health.
Correlation between quality of life changes and clinical response to growth hormone therapy | Day 0
  Correlation between the changes in scores on the 2 questionnaires QoLISSY and PedsQL 4.0 at adult size and number of centimeters taken since the start of growth hormone treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Polak, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No